CLINICAL TRIAL: NCT00002675
Title: A TRIAL OF ADJUVANT CHEMOTHERAPY IN PATIENTS WITH INTRAOCULAR RETINOBLASTOMA
Brief Title: Chemotherapy in Treating Patients With Retinoblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 95-040; CDR0000064317 (Registry Identifier: PDQ (Physician Data Query)); NCI-V95-0710
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Retinoblastoma
Keywords: intraocular retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Filgrastim; Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Mesna; Vincristine

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: mesna
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with retinoblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the response rate to adjuvant carboplatin (CBDCA) alone in children with intraocular retinoblastoma. II. Assess the overall survival, disease-free survival, and time to treatment failure in these patients. III. Attempt to maintain a 90% disease-free survival rate with this treatment. IV. Estimate the percentage of disease-free survivors who do not require the use of radiotherapy after adjuvant CBDCA. V. Assess the toxicity of this treatment. VI. Estimate the percentage of functional eyes salvaged using this radiation-sparing protocol and compare these results, in a nonrandomized manner, with historical treatment results in this population.

OUTLINE: Patients are stratified according to vitreous disease (yes vs no). Patients receive carboplatin IV over 1 hour on day 0. Treatment repeats every 2-3 weeks for 2 courses. Patients achieving complete response (CR) proceed to local control measures consisting of cryotherapy, laser photocoagulation, etc. (except brachytherapy). Patients not achieving CR continue with carboplatin until local control measures feasible. Patients with vitreous disease achieving CR receive 2 additional courses and then receive local control measures. Patients with vitreous disease not achieving CR receive intensive chemotherapy. Patients receive intensive chemotherapy consisting of vincristine IV on days 0, 7, and 14, cisplatin IV over 6 hours on day 0, etoposide IV on days 1 and 2, followed by cyclophosphamide IV over 60 minutes on days 1 and 2. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 3 and until blood counts recover. Treatment repeats every 2-4 weeks for 2 courses beyond CR. Patients are followed for 3 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study over 5-6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Intraocular retinoblastoma Ophthalmologic exam under anesthesia within 3 weeks prior to registration No pathologic confirmation required No evidence of extraocular disease, i.e.: Negative head MRI or CT (contrast not required) Negative CSF cytology Negative bone marrow aspiration and biopsy

PATIENT CHARACTERISTICS: Age: Under 18 Performance status: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 2.0 mg/dl SGOT or SGPT less than 5 times upper limit of normal Renal: Creatinine normal for age OR Creatinine clearance greater than 50 ml/min

PRIOR CONCURRENT THERAPY: No prior chemotherapy or radiotherapy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 1995-05; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States